CLINICAL TRIAL: NCT02934100
Title: Evaluation of Effectiveness of Selected Physical and Kinesiotherapeutic Methods in Patients With Lower Calcaneal Spur
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Lodz (Other)
Responsible Party: Principal Investigator, Natalia Kociuga, Master of Physical Therapy, Medical University of Lodz
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: RNN/47/16/KE
Record Dates: First submitted 2016-10-11; First posted 2016-10-14 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2016-10

CONDITIONS: Heel Spur; Calcaneal Spur
Keywords: Calcaneal spur; Heel spur; ESWT; Extracorporeal shock wave therapy; ultrasound therapy; electric field diathermy; skanlab 25 bodywave; sham laser therapy
MeSH Terms: conditions — Heel Spur

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group 1 - ESWT Treatment (Active Comparator): Patients treated with Extracorporeal Shock Wave Therapy once a week for 10 weeks
  Interventions: Device: Shock Master 300
- Group 2 - Body Wave (Active Comparator): Patients treated with electric field diathermy three times a week for 5 weeks
  Interventions: Device: Skanlab 25 BODYWAVE
- Group 3 - Ultrasound (Active Comparator): Patients treated with ultrasound therapy three times a week for 5 weeks
  Interventions: Device: EVO US13 CosmoGamma
- Group 4 - Control group (Sham Comparator): Patients treated with sham laser therapy three times a week for 5 weeks
  Interventions: Device: Sham LASER CTL1106MX

INTERVENTIONS:
Device: Shock Master 300 — Extracorporeal Shock Wave Therapy
  In all treatments (from 1 to 10) applied number of pulses is 4500 and the frequency is based on the patients feelings (from 8 to 12 Hz). Variable is the pressure:
  Treatment 1 - 2,5 Bar; Treatment 2 - 2,6 Bar; Treatment 3 - 2,7 Bar; Treatment 4 - 2,8 Bar; Treatment 5 - 3,0 Bar; Treatment 6 - 3,2 Bar; Treatment 7 - 3,4 Bar; Treatment 8 - 3,6 Bar; Treatment 9 - 3,8 Bar; Treatment 10 - 4,0 Bar.
  Each patient will also receive kinesiotherapy treatment that will consist of:
  * eight-minute massage of posterior lower leg muscles
  * plantar aponeurosis stretching
  Other Names: produced by GYMNA
  Arms: Group 1 - ESWT Treatment
Device: Skanlab 25 BODYWAVE — Electric field diathermy therapy - Capacitive energy transfer system (CETS)
  Time of each treatment (from 1 to 15) is eight minutes. Variable is the energy:
  Treatment 1 - 3; Treatment 2 - 3; Treatment 3 - 4; Treatment 4 - 4; Treatment 5 - 5; Treatment 6 - 5; Treatment 7 - 6; Treatment 8 - 6; Treatment 9 - 7; Treatment 10 - 7; Treatment 11 - 7; Treatment 12 - 7; Treatment 13 - 7; Treatment 14 - 7; Treatment 15 - 7.
  Each patient will also receive kinesiotherapy treatment that will consist of:
  * eight-minute massage of posterior lower leg muscles
  * plantar aponeurosis stretching
  Other Names: produced by SKANLAB AS
  Arms: Group 2 - Body Wave
Device: EVO US13 CosmoGamma — Ultrasound therapy
  Doses applied as following:
  Each treatment (from 1 to 15) is pulsed ultrasound (1MHz, pulsed 1:4). Variable is the time and intensity:
  Treatment 1 - 4 minutes, 0,4 W/cm2; Treatment 2 - 5 minutes, 0,4 W/cm2; Treatment 3 - 5 minutes, 0,5 W/cm2; Treatment 4 - 6 minutes, 0,5 W/cm2; Treatment 5 - 6 minutes, 0,6 W/cm2; Treatment 6 - 6 minutes, 0,6 W/cm2; Treatment 7 - 6 minutes, 0,6 W/cm2; Treatment 8 - 6 minutes, 0,7 W/cm2; Treatment 9 - 7 minutes, 0,7 W/cm2; Treatment 10 - 7 minutes, 0,7 W/cm2; Treatment 11 - 7 minutes, 0,8 W/cm2; Treatment 12 - 8 minutes, 0,8 W/cm2; Treatment 13 - 8 minutes, 0,8 W/cm2; Treatment 14 - 8 minutes, 0,8 W/cm2; Treatment 15 - 8 minutes, 0,8 W/cm2.
  Each patient will also receive kinesiotherapy treatment that will consist of:
  * eight-minute massage of posterior lower leg muscles
  * plantar aponeurosis stretching
  Other Names: produced by EMILDUE
  Arms: Group 3 - Ultrasound
Device: Sham LASER CTL1106MX — Sham laser therapy Time of each treatment (from 1 to 15) is four to five minutes. Developed is 10 points, each point takes 15 seconds. Device is unplugged and it does not emit any radiation.The patient does not know that the procedure is not really executed.
  Each patient will also receive kinesiotherapy treatment that will consist of:
  * eight-minute massage of posterior lower leg muscles
  * plantar aponeurosis stretching
  Other Names: produced by CTL
  Arms: Group 4 - Control group

SUMMARY:
This study evaluates the effectiveness of physiotherapy and kinesiotherapy in patients with calcaneal spurs. the aim of the study is to compare the efficacy of calcaneal spurs treatment provided with extracorporeal shock wave therapy, ultrasound therapy, electric field diathermy associated with kinesiotherapy and sham laser in combination with kinesiotherapy. In each group kinesiotherapy treatment is the same and consists of an eight-minute massage of posterior lower leg muscles and plantar aponeurosis stretching.

DETAILED DESCRIPTION:
Number of 120 diagnosed with heel spur patients, will be allocated randomly into one of three treatment groups or into the control group. Assignment to a group is random, but before that happens patients will be questioned about inclusion and exclusion criteria of the study. Depending on group allocation, patients in treatment groups will receive one of the following physical therapy treatments:

* ESWT (once a week for 10 weeks)
* ultrasound (three times a week for 5 weeks)
* electric field diathermy (three times a week for 5 weeks).

Patients allocated in control group, will receive a sham laser therapy (only the timer on the machine activated) three times a week for 5 weeks.

Regardless of affiliation to the group, each patient will also receive kinesiotherapy treatment.

At the beginning of the study, each patient receives the "Information for the patient," describing the exact course of each stage of the study, then signs a "Form of informed consent to participate in the study.". The next stage of the study is to fill in the participant survey questionnaire and physical examination provided by the researcher.

Assessment of improvements will be made twice: right after the therapy and two months later. Every stage of the study is carried out by one and the same investigator.

ELIGIBILITY:
Inclusion Criteria:

* heel spur (calcaneal spur) diagnosed by a doctor based on X-ray examination, diagnostic ultrasonography or MR
* signed informed consent
* heel pain for at least one month

Exclusion Criteria:

* pregnancy
* generalized acute infection (fever, cough, runny nose)
* local infection in the treated leg (wound, swelling)
* cancer
* injections of corticosteroids in the last six weeks
* pacemaker
* acute inflammation of the joints of the lower limbs
* inflammation of the veins
* Fresh fractures, post-traumatic
* osteoporosis
* Reynaud's disease
* Burger disease
* atherosclerosis
* after surgery condition before removing stitches
* High blood pressure
* after CT with contrast condition in the last two weeks
* The state of the lumbar puncture
* Strong imbalance
* Condition after myocardial infarction in the last six weeks
* Rheumatoid arthritis
* Ankylosing spondylitis
* Significant leg ulcers
* diabetes
* The risk of bleeding in the muscle tissue
* Thromboangiitis
* Hypersensitivity skin in the treated section
* A tendency to hemorrhage
* Pathological arrogance bone under the skin in the treated section
* Metal implants and surgical implants in the area of the lower limb subjected to therapy

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-08; Primary Completion 2017-08 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
The American Orthopedic Foot and Ankle Society Score (AOFAS) - Change | Change from before the treatment and right after the treatment. Also change from after the treatment at 2 months.
  The American Orthopedic Foot and Ankle Society Score (AOFAS) is one of most widely used clinician-reporting tools for foot and ankle conditions. Developed in 1994, it is a clinician-based score that measures outcomes for four different anatomic regions of the foot: The ankle-hindfoot, midfoot, metatarsophalangeal (MTP)-interphalangeal (IP) for the hallux, and MTP-IP for the lesser toes.
  The four anatomic regions of the AOFAS are all represented by a different version of the survey with each tool designed to be used independently. The questionnaire consists of nine items that are distributed over three categories: Pain (40 points), function (50 points) and alignment (10 points). These are all scored together for a total of 100 points.
The SF-36v2 Health Survey (SF-36v2) - Change | Change from before the treatment and right after the treatment. Also change from after the treatment at 2 months.
  The SF-36v2 Health Survey is a multipurpose, short-form health survey with 36 questions that yields an eight-scale profile of functional health and well-being, as well as two psychometrically based physical and mental health summary measures and a preference-based health utility index. Like its predecessor, the SF-36 Health Survey , the SF-36v2 is a generic measure of health status, as opposed to one that targets a specific age, disease, or treatment group. It has proven useful for conducting surveys of general and specific populations, comparing the relative burden of diseases, and differentiating the health benefits produced by a wide range of treatments.
The Laitinen Pain Indicator Questionnaire | Change from before the treatment and right after the treatment. Also change from after the treatment at 2 months.
  The Laitinen Pain Indicator Questionnaire is subjective and point tool which is used to assess the level of pain. Patients have to evaluate four indicators: pain intensity, the frequency of pain, the frequency of use of analgesics and physical activity limitations. Each indicator score is assigned from 0 to 4, with 0 being no problem, and four being a maximum problem.

SECONDARY OUTCOMES:
Two weights test | Patients will be screened using this scale three times: before treatment, immediately after its completion and two months after the end of therapy.
  The two weights test is measures the uniformity of the load of the lower limbs. The patient gets the right lower limb on one scale and another limb on the other scale. By standing on the scales must look ahead. The range of measurement error is five kilograms.
Heel standing test | Patients will be screened using this scale three times: before treatment, immediately after its completion and two months after the end of therapy.
  The heel standing test is to measure the intensity of pain experienced by burdening calcaneus. The patient is standing by the wall and must stand on both heel bones at the same time, then turn on the right calcaneus and then on the left calcaneus. Each of the three above mentioned activities is assessed using a three-point scale, depending on the feasibility of the task by the patient: job done at 100-75% without much problem, the task done at 75-25% with difficulty, the task done at 25-0% with great difficulty, or not done at all.
  The test was created for this study and a researcher authorship.
The Visual Analogue Scale | Patients will be screened using this scale three times: before treatment, immediately after its completion and two months after the end of therapy.
  The visual analogue scale is a measurement instrument that is used for subjective assessment of pain made by the patient. The pain can be evaluated in a ten-point scale, where one represents no pain and ten is the pain unbearable.

CONTACTS AND LOCATIONS:
Overall Officials: Natalia Kociuga, master, Principal Investigator — Medical University of Lodz, Poland
Locations (1):
- Non-public health care facility "NZOZ Komed", Lodz, Łódź Voivodeship, Poland

REFERENCES:
- See also: review article describing what the "heel spurs" really are and what are their consequences — http://czyrny.pl/pdf/Art_01_czyrny.JOTSRR.2.2010.pdf